CLINICAL TRIAL: NCT01108497
Title: Genome, Proteome and Tissue Microarray in Childhood Acute Leukemia
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSHEM0001; 11062 (Other: Stanford IRB); SU-09112009-3881 (Other: Stanford University)
Record Dates: First submitted 2010-04-20; First posted 2010-04-22 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow

INTERVENTIONS:
Procedure: Bone Marrow Aspiration

SUMMARY:
We will study gene and protein expression in leukemia cells of children diagnosed with acute leukemia. We hope to identify genes or proteins which can help us grade leukemia at diagnosis in order to: (a) develop better means of diagnosis and (b) more accurately choose the best therapy for each patient.

ELIGIBILITY:
Inclusion Criteria:1. All children who present at Packard hospital with a new diagnosis or relapse of acute leukemia will be eligible. There is no bias in regards to age range, gender or ethnic background.

2. Signed informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children who present at Packard hospital with a new diagnosis or relapse of acute leukemia will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2001-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Gene Expression | days 0, 8, 22 or 29

CONTACTS AND LOCATIONS:
Overall Officials: Norman James Lacayo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States